CLINICAL TRIAL: NCT06969690
Title: Question-Order Effect Experiment to Measure HIV Stigma Among Persons With HIV (PWH) in Rural Uganda
Brief Title: Question-Order Effect Experiment to Measure HIV Stigma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Mbarara University of Science and Technology (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Alexander Tsai, Associate Professor of Psychiatry, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2013P000395_5; R01MH125667 (NIH)
Record Dates: First submitted 2025-05-05; First posted 2025-05-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: HIV
Keywords: HIV stigma; discrimination

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- V1 (Experimental): As this is a survey experiment, the "intervention" involves random assignment to a survey questionnaire with specific treatments. The first treatment is a questionnaire with questions about internalized stigma followed by questions of experienced stigma. Each question is answered as Yes/No/It depends on knowing more details.
  Interventions: Other: Survey questionnaire V1
- V2 (Experimental): As this is a survey experiment, the "intervention" involves random assignment to a survey questionnaire with specific treatments. The second treatment is a questionnaire with questions about experienced stigma followed by questions about internalized stigma. Each question is answered as Yes/No/It depends on knowing more details.
  Interventions: Other: Survey questionnaire V2

INTERVENTIONS:
Other: Survey questionnaire V1 — Each version of the questionnaire includes a different order of statements about which study participants are asked to provide a Yes, No, or It depends response.
  Arms: V1
Other: Survey questionnaire V2 — Each version of the questionnaire includes a different order of statements about which study participants are asked to provide a Yes, No, or It depends response.
  Arms: V2

SUMMARY:
Question-order effect experiment to measure HIV-related stigma among people living with HIV (PWH).

DETAILED DESCRIPTION:
HIV-related stigma is a barrier to engagement in HIV prevention and treatment. Given the negative impact of stigma on the HIV continuum of care, accurate assessment of HIV-related stigma among people living with HIV (PWH) in resource-limited settings is paramount. The purpose of this study is to conduct a question order experiment to assess the extent to which the order of presented questions affects measurement of HIV-related stigma.

ELIGIBILITY:
Inclusion Criteria:

- All HIV-positive (self-reported) adults who consider Nyakabare their primary place of residence and who are capable of providing consent

Exclusion Criteria:

* Minors younger than 18 years of age, with the exception of emancipated minors
* Persons who do not consider Nyakabare Parish their primary place of residence, e.g. persons who happen to be visiting Nyakabare at the time of the survey or who own a home in Nyakabare but spend most of their time outside of the parish
* Persons with psychosis, neurological damage, acute intoxication, or other cognitive impairment (all of which are determined informally in the field by non-clinical research staff in consultation with a supervisor)
* Persons who are not HIV positive

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2023-11-02 (Actual); Primary Completion 2025-01-06 (Actual); Study Completion 2025-01-06 (Actual)

PRIMARY OUTCOMES:
Self-esteem | Baseline (assessed at the time the survey is administered)
  ...do you think less of yourself because of your HIV status? (single item)
Self-respect | Baseline (assessed at the time the survey is administered)
  ...have you felt ashamed because of your HIV status? (single item)
Experiences of harassment due to HV status | Baseline (assessed at the time the survey is administered)
  * have you lost respect or standing in the community because of your HIV status?
  * have people talked badly about you because of your HIV status?
  * have you been verbally insulted, harassed and/or threatened because of your HIV status?
  * have you been physically assaulted because of your HIV status?
  * has someone else disclosed your HIV status without your permission?
  * have you felt that people have not wanted to sit next to you, for example on public transport, at church or in the waiting room, because of your HIV status? (six items)

CONTACTS AND LOCATIONS:
Overall Officials: Alexander C Tsai, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Mbarara University of Science and Technology, Mbarara, Uganda

IPD SHARING:
Plan to Share IPD: No